CLINICAL TRIAL: NCT00985842
Title: Socket System Effect on Tissue Oxygenation During Amputee Gait
Brief Title: Study to Determine if Different Prosthetic Sockets Effect How Much Oxygen is in the Tissue of Lower Limb Amputees While They Are Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A4378-R
Record Dates: First submitted 2007-12-11; First posted 2009-09-29 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Amputation; Diabetes Complications; Leg Injuries; Traumatic Amputation
Keywords: Artificial limbs; Gait; Oximetry; Prosthesis; Rehabilitation
MeSH Terms: conditions — Diabetes Complications; Leg Injuries; Amputation, Traumatic | interventions — Suction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Other): Comparison of five different clinically used suspension and socket systems
  Interventions: Device: Pe-Lite and sleeve suspension socket; Device: Total Surface bearing a socket with a sleeve suspension but without suction; Device: Total surface bearing suction socket with a pin lock suspension; Device: Total surface bearing suction socket with a sleeve suspension; Device: Vacuum-assisted socket system (Harmony System, Otto Bock)

INTERVENTIONS:
Device: Pe-Lite and sleeve suspension socket — Prosthetic socket worn by the amputee that has a Pe-lite foam liner between the socket and the residual limb. It is suspended from the residual limb using a sleeve at the top of the socket.
Device: Total Surface bearing a socket with a sleeve suspension but without suction — Prosthetic socket worn by the amputee where the fit of the socket touches every part of the residual limb. This socket is suspended from the residual limb using a sleeve at the top of the socket.
Device: Total surface bearing suction socket with a pin lock suspension — Prosthetic socket worn by the amputee where the fit of the socket touches every part of the residual limb. This socket is suspended from the residual limb using a pin that protrudes from the bottom of the liner into the socket that is then locked in place by the amputee.
Device: Total surface bearing suction socket with a sleeve suspension — Prosthetic socket worn by the amputee where the fit of the socket touches every part of the residual limb. This socket using vacuum suction plus a sleeve at the top of the prosthetic socket to enhance the security of the suspension.
Device: Vacuum-assisted socket system (Harmony System, Otto Bock) — Prosthetic socket worn by the amputee where the a vacuum pump, in this case a mechanically-activated pump, creates a vacuum between the socket and the limb. This vacuum suspends the prosthetic limb from the amputee's residual limb.

SUMMARY:
Amputee gait produces periodic occlusion of residual limb blood vessels. During the stance phase of gait, body weight cause the prosthesis to compresses the soft tissue of the residual limb and occlude blood flow. This occlusion can be relieved during swing phase, but may depend on type of prosthesis. The purpose of the proposed research is to: (1) discover the range of tissue oxygenation in the intact and residual lower limbs of dysvascular amputees during gait and (2) to learn which of five different prosthetic limb systems provides greater tissue oxygenation.

DETAILED DESCRIPTION:
The amount of oxygen in residual limb tissue is an important health status indicator; resistance to infection, promotion of wound healing, production of collagen, and epithelialization all correlate with higher oxygen levels. Unfortunately, simply donning a lower limb prosthesis may limit circulation and reduce the level of tissue oxygenation. This reduction may be compounded by the biomechanical forces of gait. The compressive loads of the body's weight during stance and the inertial loads of the prosthesis during swing may further occlude circulation, albeit by different mechanisms.

For the dysvascular lower limb amputee, the choice of prosthetic socket and suspension system may impact the overall health of their residual limb and wound healing capacity. An inappropriate choice may lead to skin irritation, tissue breakdown, discomfort, and reduced mobility. For these patients, any component that reduces tissue oxygenation is a significant problem because compromised circulation can forestall wound healing.

The objective of the proposed research is to use photo-oximetry to discover which of five different prosthetic limb systems results in higher residual limb tissue oxygenation during both rest and gait. This experiment will enable evidence-based decision making on this clinically relevant problem. Using a prospective, randomized cross-over experimental design and the investigators' photo-oximetry system, the investigators will measure and compare the tissue oxygenation along the medial and lateral surfaces (3 sites each) of the residual limb during rest and walking.

ELIGIBILITY:
Inclusion Criteria:

All subjects must meet the following inclusion criteria:

* unilateral transtibial amputee of diabetic etiology between the ages of 18 and 70,
* have been fit with a prosthesis and have used a prosthesis for at least one year,
* wear the prosthesis at least 4 hours per day,
* ambulate without upper extremity aids, and
* have no history of injurious falls within the previous six months.

Exclusion Criteria:

Subjects will be excluded if:

* they have a significant lower extremity pain condition, musculoskeletal disorder, or neurological deficit that interferes with their ability to pursue typical daily activities or alters their gait characteristics or
* their residual limb is ulcerated.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-11-01 (Actual); Primary Completion 2012-10-26 (Actual); Study Completion 2012-10-26 (Actual)

PRIMARY OUTCOMES:
Oxygen in tissue | Comparison of five different systems will be performed in one session occurring on one day
  Tissue oxygen saturation (StO2)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn K Klute, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information about this study: Socket System Effect on Tissue Oxygenation During Amputee Gait — http://www.amputation.research.va.gov/